CLINICAL TRIAL: NCT03875534
Title: ACHieve: A Multi-center, Longitudinal, Observational Study of Children With Achondroplasia
Brief Title: A Multi-center, Longitudinal, Observational Study of Children With Achondroplasia
Status: Completed | Type: Observational
Sponsor: Ascendis Pharma A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: TCC-NHS-01
Record Dates: First submitted 2019-03-07; First posted 2019-03-14 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Achondroplasia
Keywords: Achondroplasia; Dwarfism
MeSH Terms: conditions — Achondroplasia; Dwarfism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a long-term, multi-center, longitudinal, observational study in children with achondroplasia (ACH). The aim is to study height velocity and comorbidities in children with ACH. This is a natural history study and no study medication will be administered.

ELIGIBILITY:
Inclusion Criteria:

1. Legally authorized representative is willing and able to provide written, signed informed consent (with a written assent from the child when appropriate per local requirements)
2. Willing and able to comply with study protocol per investigator judgement
3. Clinical diagnosis of achondroplasia (confirmed by the investigator)
4. Age between 0 to 8 years old at enrollment
5. Able to stand without assistance (if the child is 24 months or older)

Exclusion Criteria:

1. Have received chronic treatment (> 3 months) of human growth hormone (hGH) or other medicinal products intended to affect stature or body proportionality at any time
2. Have received any dose of medicinal products intended to affect stature or body proportionality within the previous 6 months of screening
3. Have received any investigational medicinal product or device intended to affect stature or body proportionality at any time
4. History or presence of injury or disease of the growth plate(s), other than ACH, that affects growth potential of long bones
5. History of any bone-related surgery that affects growth potential of long bones, such as orthopedic reconstructive surgery and osteotomy (foramen magnum decompression, and laminectomy with full recovery are allowed with minimum of 6 months of bone healing. Limb-lengthening with full recovery is allowed with a minimum of 12 months of bone healing.)
6. Have forms of skeletal dysplasias other than achondroplasia or medical conditions that result in short stature or abnormal bone growth [such as severe achondroplasia with developmental delay and acanthosis nigricans (SADDAN), hypochondroplasia, growth hormone deficiency, Turner syndrome, pseudoachondroplasia. uncontrolled hypothyroidism, uncontrolled diabetes mellitus, autoimmune disease requiring corticosteroid therapy, inflammatory bowel disease, and chronic renal insufficiency]
7. History or presence of malignant disease, other than basal cell epithelioma/carcinoma or completely resected squamous skin cancer with no recurrence for 12 months per medical records

Ages: 0 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants and children with achondroplasia from birth to 8 years of age.
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Annualized height velocity (centimeters/year) in children with achondroplasia | Up to 5 years
  Subjects will undergo a series of height measurements (in centimeters) on Day 1 and then every 6 months over the study period with height velocity reported in cm/year

SECONDARY OUTCOMES:
Collection of natural history of achondroplasia symptoms in children with achondroplasia | Up to 5 years
  To characterize achondroplasia symptoms in children with achondroplasia

CONTACTS AND LOCATIONS:
Locations (35):
- United States (10):
  - Ascendis Pharma Investigational Site, Little Rock, Arkansas
  - Ascendis Pharma Investigational Site, Oakland, California
  - Ascendis Pharma Investigational Site, Aurora, Colorado
  - Ascendis Pharma Investigational Site, Wilmington, Delaware
  - Ascendis Pharma Investigational Site, Saint Paul, Minnesota
  - Ascendis Pharma Investigational Site, Columbia, Missouri
  - Ascendis Pharma Investigational Site, Buffalo, New York
  - Ascendis Pharma Investigational Site, Houston, Texas
  - Ascendis Pharma Investigational Site, Seattle, Washington
  - Ascendis Pharma Investigational Site, Madison, Wisconsin
- Ascendis Pharma Investigational Site, Parkville, Victoria, Australia
- Ascendis Pharma Investigational Site, Linz, Austria
- Canada (3):
  - Ascendis Pharma Investigational Site, Edmonton, Alberta
  - Ascendis Pharma Investigational Site, Ottawa, Ontario
  - Ascendis Pharma Investigational Site, Montreal, Quebec
- China (6):
  - Ascendis Pharma Investigational Site, Beijing
  - Ascendis Pharma Investigational Site, Guangzhou
  - Ascendis Pharma Investigational Site, Hangzhou
  - Ascendis Pharma Investigational Site, Shanghai
  - Ascendis Pharma Investigational Site, Shenzhen
  - Ascendis Pharma Investigational Site, Wuhan
- Ascendis Pharma Investigational Site, Copenhagen, Capital Region, Denmark
- Ascendis Pharma Investigational Site, Paris, France
- Ascendis Pharma Investigational Site, Berlin, Germany
- Ascendis Pharma Investigational Site, Dublin, Ireland
- Ascendis Pharma Investigational Site, Milan, Italy
- Ascendis Pharma Investigational Site, Auckland, New Zealand
- Ascendis Pharma Investigational Site, Coimbra, Portugal
- Spain (4):
  - Ascendis Pharma Investigational Site, Barcelona
  - Ascendis Pharma Investigational Site, Esplugues de Llobregat
  - Ascendis Pharma Investigational Site, Madrid
  - Ascendis Pharma Investigational Site, Vitoria-Gasteiz
- Ascendis Pharma Investigational Site, Lausanne, Switzerland
- United Kingdom (2):
  - Ascendis Pharma Investigational Site, Glasgow
  - Ascendis Pharma Investigational Site, London

IPD SHARING:
Plan to Share IPD: No